CLINICAL TRIAL: NCT04628338
Title: A Pilot Study of IFN-γ to Treat Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) That Has Relapsed After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: IFN-γ to Treat Acute Myeloid Leukemia (AML) and Myelodysplastic Syndrome (MDS) That Has Relapsed After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sawa Ito, MD (Other)
Collaborators: Horizon Pharma USA, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Sawa Ito, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 20-092
Record Dates: First submitted 2020-10-29; First posted 2020-11-13 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Myelodysplastic Syndromes; Myeloid Leukemia; Allogeneic Stem Cell Transplantation
Keywords: allogeneic hematopoietic stem cell transplantation; acute myeloid leukemia; myelodysplastic syndrome; graft versus host disease; AML; MDS; alloSCT; GVHD; interferon-gamma-1b; Actimmune; IFN-g; donor lymphocyte infusion
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid; Leukemia, Myeloid, Acute; Graft vs Host Disease | interventions — interferon gamma-1b; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IFN-γ (Experimental): 100mcg IFN-γ subcutaneously three times per week (Weeks 0-7), once per week (Weeks 8-12) (or per protocol guidance based on tolerability, response, or DLI infusions)
  Interventions: Drug: IFN-γ (interferon gamma-1b) injection

INTERVENTIONS:
Drug: IFN-γ (interferon gamma-1b) injection — Dosage form: 100 mcg (2 million International Units) per 0.5 mL solution, administered subcutaneously Dose regimen: three times weekly (Weeks 0-7), once weekly (Weeks 8-12)
  Other Names: ACTIMMUNE®

SUMMARY:
This study proposes a safe dosing regimen IFN-γ that is sufficient to stimulate IFN-γ receptors on malignant blasts in patients who developed relapsed acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) after alloSCT with no active or history of III-IV acute graft-versus-host disease (GVHD). It is hypothesized that IFN-γ will promote graft-vs-leukemia (GVL) in patients with AML/MDS that has relapsed after alloSCT.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (alloSCT) can cure patients with acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). However, relapsed AML/MDS is the most significant single cause of treatment failure, and the majority of relapsed patients ultimately succumb. Alloreactive T cells in the donor graft can kill residual leukemia cells, mediating the graft-vs-leukemia (GVL) effect. Consistent with this, recipients of T cell-depleted grafts have higher rates of relapse. GVL is more potent against chronic leukemias than acute myeloblastic diseases, and the higher incidence of relapse in patients with AML/MDS reflects a failure in GVL.

The central goal of this pilot trial will be to explore whether IFN-γ in this setting is safe and whether it has the desired biological activities on malignant blasts in vivo. IFN-γ will be tested in relapsed patients as monotherapy and in conjunction with donor leukocyte infusions (DLI). The clinical and biological information from this study is essential to design a phase II trial with a therapeutic endpoint.

Treatment will be initiated at 100mcg (almost equal to the dose of 50 mcg/m2 for an adult) three times a week, with the potential to deescalate the frequency of injection for unacceptable toxicity. To explore whether this dosing regimen is sufficient to activate myeloblasts, pre- and post-treatment bone marrow specimens will be harvested to analyze for IFN-γ action (upregulation of HLA class I; HLA class II, ICAM-1 and phosphorylation of STAT1). The primary safety concern is the development of GVHD, which is routinely monitored for all alloSCT patients.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of allogeneic stem cell transplantation for acute myeloid leukemia or myelodysplastic syndrome from a human leukocyte antigen (HLA) matched donor
* Relapsed of primary disease with 5% to 20% of blasts in the bone marrow by flow cytometry in the bone marrow with an clear leukemia-associated immunophenotype (If the patient received therapy to treat the relapse, he or she must have 5-20% residual blasts prior to enrollment on this study)
* Performance status KPS score >60% (ECOG 0-2)
* No increases in systemic immunosuppression in the prior four weeks other than to maintain therapeutic levels
* No systemic corticosteroid with a dose higher than 0.5mg/kg/day prednisone or equivalent
* No history of grade IV acute GVHD
* No new systemic immunosuppressive medications in the prior two weeks initiated due to GVHD
* Willingness to have bone marrow and peripheral blood collected as per the study protocol
* Must be able to give informed consent
* Age 18 or older

Exclusion Criteria:

* Contraindication to receive IFN-γ including known hypersensitivity to interferon-gamma, E. coli derived products or any component of the product
* Subjects with a positive pregnancy test or who are breastfeeding
* For men or women of childing bearing potential (age < 50 without hysterectomy or oophorectomy or documented menopause), unwilling to use effective contraception for the duration of the study.
* Primary engraftment failure
* Active cardiac arrhythmias not controlled by medical management or current NYHA class II or higher congestive heart failure
* Active ischemic heart disease not well controlled with medications
* A seizure disorder not well controlled by medications
* Estimated GFR <30 mL/min
* AST/SGOT or ALT/SPOT > 5 x ULN
* Total bilirubin > 3 x ULN
* Chemotherapy (other than hypomethylating and/or venetoclax therapy) within the prior 4 weeks
* Body surface area at or less than 1.5 m2, or greater than 2.5 m2 so as to minimize the variation in IFN-γ exposure based on differences in BSA.
* Patients less than 18 years old.
* Pregnant or breastfeeding patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Upregulation HLA l (HLA-ABC) | Up to 6 months
  Upregulation of HLA l (HLA-ABC) in bone marrow malignant blasts post-IFN-γ treatment, measured by the change in mean florescent intensity by flow cytometry.
Upregulation of HLA ll (HLA-DR/DQ) | Up to 6 months
  Upregulation of HLA ll (HLA-DR/DQ) in bone marrow malignant blasts post-IFN-γ treatment, measured by the change in mean florescent intensity by flow cytometry.
Upregulation of ICAM-1 | Up to 6 months
  Upregulation of ICAM-1 in bone marrow malignant blasts post-IFN-γ treatment, measured by the change in mean florescent intensity by flow cytometry as a percentage of positive cells.
Adverse events related to IFN-γ | Up to 6 months
  Adverse events of IFN-γ in relapsed patients after alloSCT per CTCAE v5.0.
Generation of phosphorylated-STAT1 | Up to 6 months
  Generation of phosphorylated-STAT1 in bone marrow malignant blasts post-IFN-γ treatment, measured by the change in mean florescent intensity by flow cytometry as a percentage of positive cells.

SECONDARY OUTCOMES:
Malignant Blast Burden | Up to 6 months
  Change in malignant blasts number after IFN-γ therapy and subsequent donor lymphocyte infusion.
Incidence of GVHD | Up to 6 months
  Incidence of Graft Versus Host Disease (GVHD) progression or de novo GVHD after INF-g therapy and subsequent donor lymphocyte infusion.
Incidence of de novo GVHD | Up to 6 months
  Incidence of graft-versus-host disease (GVHD) progression after IFN-γ therapy and subsequent DLI.

CONTACTS AND LOCATIONS:
Overall Officials: Sawa Ito, MD; PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ito S, Geramita E, Ventura K, Neupane B, Bhise S, Moore EM, Furlan S, Shlomchik WD. IFN-gamma and donor leukocyte infusions for relapsed myeloblastic malignancies after allogeneic hematopoietic stem cell transplantation. JCI Insight. 2025 Mar 25;10(9):e190655. doi: 10.1172/jci.insight.190655. eCollection 2025 May 8. PMID 40131369
- See also: IFN-γand donor leukocyte infusions for relapsed myeloblastic malignancies after allogeneic hematopoietic stem cell transplantation - PubMed — https://pubmed.ncbi.nlm.nih.gov/40131369/